CLINICAL TRIAL: NCT00063310
Title: Antigonadotropin-Leuprolide in Alzheimer's Disease Drug INvestigation (ALADDIN)
Brief Title: ALADDIN Study: Antigonadotropin-Leuprolide in Alzheimer's Disease Drug INvestigation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Voyager Pharmaceutical Corporation (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0047; IND 66,415
Record Dates: First submitted 2003-06-25; First posted 2003-06-26 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Aging Women; Hormone therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Leuprolide

INTERVENTIONS:
Drug: Leuprolide acetate

SUMMARY:
ALADDIN is a research study to investigate the safety and effectiveness of leuprolide (a hormone drug) to improve the cognitive function and slow the progression of Alzheimer's disease (AD). In women leuprolide is commonly used to treat hormone related conditions such as endometriosis and uterine fibroids. The study will include treatment of women 65 years and older with mild to moderate Alzheimer's disease who reside in the community.

DETAILED DESCRIPTION:
The study will include the treatment of participants with mild to moderate AD, and the objective is to evaluate the safety and efficacy of two different doses of leuprolide to improve the cognitive function and slow the progression of AD, as measured by the ADAS-COG and the Clinical Global Impression (CGI). Measures of behavioral disturbances and quality of life of the caregiver will be made also. The study design is randomized, double blind, placebo-controlled, parallel group design with a 2:1 randomization of drug to placebo. Sample size will include 90 participants

ELIGIBILITY:
Inclusion Criteria:

Patients who satisfy all of the inclusion criteria listed below will be eligible for entry into the trial. Patients will be considered eligible if:

* They give their consent by signing the IRB-approved Informed Consent Form and the responsible caregiver also signs the consent form; or, if the patient is judged by the Investigator to be unable to give consent, if the legally authorized representative gives consent by signing the consent form and the patient gives assent, in accord with local regulations;
* They are female;
* They are 65 years of age or older;
* They have a diagnosis of probable AD according to the National Institute of Neurological Disorders-Alzheimer's Disease and Related Disorders Association (NINDS-ADRDA) criteria and the Investigator ascertains that the condition was present at least 6 months prior to screening;
* They are taking a cholinesterase inhibitor, they began taking it at least 90 days prior to baseline and, in the Investigator's opinion, the dosage will likely remain stable throughout the trial;
* They are taking other drugs or substances that have purported cognition enhancing properties such as ginkgo biloba and Vitamin E, they began taking it at least 60 days prior to baseline and, in the Investigator's opinion, the dosage will likely remain stable throughout the trial;
* They score no lower than 12 or higher than 24 on the (MMSE) administered at the screening visit;
* They have had a brain imaging study (CT scan, MRI or PET) performed at the time of their initial diagnosis of AD or after that time, and the findings were consistent with a diagnosis of probable AD, or, if a brain imaging study has not been performed, one will be performed during the screening process;
* Their Rosen Modified Hachinski score was 4 or lower at the screening visit, supporting the Investigator's clinical judgment that the patient's dementia is probable AD and not of vascular origin;
* They are fluent in English or Spanish and completed at least 6 years of education;
* They live at home or in a congregate living facility for requirements other than skilled nursing care, and have a caregiver who sees the patient at least three time a week for a total of at least 10 hours and can sign the consent form, provide information pertinent to the patient's cognitive status, accompany the patient on clinic visits and participate in the evaluations;
* Their hormone replacement therapy (HRT), if any, has been stable for at least 60 days prior to baseline, and is not expected to change during the course of the trial;
* They score less than 15 on the Hamilton Depression Scale (17-item version) (HamD) administered as part of the screening evaluation;
* Absorptiometry (dual-energy x-ray absorpometry (DEXA) scan), performed at screening, was within normal limits (i.e., a T- score of no less than -2.0); or, if their DEXA measure was abnormally low, they were receiving treatment for osteoporosis for at least 3 weeks and that treatment is not expected to change during the course of the trial; or, if their DEXA measure was abnormally low and they are not receiving treatment for osteoporosis, they may enter the trial after 3 weeks of treatment provided that assessments of the HamD, concomitant medications, ECG tracing and laboratory tests performed within 45 days of baseline show that they are eligible.
* values on their screening laboratory tests do not indicate significant medical conditions that would interfere with their participation in and completion of the study

Exclusion Criteria:

Patients with any of the exclusion criteria listed below will be ineligible for entry into the study. Patients will be declared ineligible if:

* They are male;
* They are younger than 65 years of age;
* They have significant neurological disease affecting the brain or psychiatric disease other than AD, such as major depression, schizophrenia, epilepsy, Parkinson's disease, or stroke;
* They have current significant systemic illness or symptoms of organ failure;
* The screening ECG shows evidence of a serious and/or unstable condition or a recent (within 6 months) myocardial infarction;
* They have a history of cancer within the last 5 years, except for basal cell or squamous cell cancer, or cervical carcinoma in situ;
* They are taking a cholinesterase inhibitor (tacrine, donepezil, rivastigmine, or galantamine) for less than 90 days prior to baseline; or, in the opinion of the Investigator, they are likely to either require a change in dose or discontinuation of the drug
* They have never received cholinesterase inhibitor treatment and are likely to initiate it;
* They started or changed within 60 days prior to the screening visit the dosage of any drug (including an over the counter drug) that affects cognitive function, such as neuroleptics, antidepressants, anxiolytics, sedatives, hypnotics, anti-convulsants, centrally acting antihypertensive agents such as clonidine and Aldomet; or other medications that have been shown to have possible effects on cognition such as Vitamin E, non steroidal anti-inflammatory drugs, statins, and hormone replacement therapy, or if, in the Investigator's opinion, the dosage of such medication is likely to be changed during the course of this trial. Any changes in the dosage of any of these drugs during the course of the trial and the reason for the change must be fully recorded in the concomitant medication page of the patient's case report form (CRF). If a drug that affects cognition is given on a PRN basis, such treatment should be interrupted for 12 hours before a visit, it at all possible;
* They are receiving coumadin or anti-Parkinsonian medications;
* They have received other investigational drugs within 30 days or 5 half-lives prior to randomization, whichever is longer;
* They are taking other medications known to affect serum gonadotropin (Gn) concentrations, such as goserelin or danazol, except for estrogen and/or progesterone;
* They have a history of bone fracture possibly secondary to low bone mass density;
* They have a history of osteoporosis not associated with bone fracture unless they are receiving therapy for osteoporosis for at least 3 weeks, and the treatment regimen is expected to stay stable their DEXA measures were abnormally low (i.e., T-score <-2.0) and they were not receiving treatment for osteoporosis for at least 3 weeks;
* They have a screening HamD score of 15 or higher;
* Their abuse or dependence on alcohol or other substances satisfy criteria for DSM-IV categories 303.9 or 305; or
* They have donated blood within 30 days of baseline or are likely to do so during the course of the trial.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90
Dates: Start 2003-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Bowen, MD, Principal Investigator — Voyager Pharmaceutical Corporation
Locations (3):
- United States (3):
  - Sun Health Research Institute, Sun City, Arizona
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Meridien Research, St. Petersburg, Florida

REFERENCES:
- [Background] Smith MA, Perry G, Atwood CS, Bowen RL. Estrogen replacement and risk of Alzheimer disease. JAMA. 2003 Mar 5;289(9):1100; author reply 1101-2. doi: 10.1001/jama.289.9.1100-a. No abstract available. PMID 12622570
- [Background] Bowen RL, Smith MA, Harris PL, Kubat Z, Martins RN, Castellani RJ, Perry G, Atwood CS. Elevated luteinizing hormone expression colocalizes with neurons vulnerable to Alzheimer's disease pathology. J Neurosci Res. 2002 Nov 1;70(3):514-8. doi: 10.1002/jnr.10452. PMID 12391612
- [Background] Short RA, Bowen RL, O'Brien PC, Graff-Radford NR. Elevated gonadotropin levels in patients with Alzheimer disease. Mayo Clin Proc. 2001 Sep;76(9):906-9. doi: 10.4065/76.9.906. PMID 11560301